CLINICAL TRIAL: NCT05427578
Title: Brain Markers of Depression Vulnerability: the Case of Prefrontal Haemodynamic Response
Status: Completed | Type: Observational
Sponsor: Dr Georg Kranz (Other)
Responsible Party: Sponsor-Investigator, Dr Georg Kranz, Principal Investigator, The Hong Kong Polytechnic University
Organization: The Hong Kong Polytechnic University (Other)
Other Study IDs: HSEARS20210323001-01
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2024-12

CONDITIONS: Depression
Keywords: remitted major depression; depression vulnerability
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Without collecting biospecimen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Remitted depression: Patients in full remission of a major depressive disorder (rMDD)
  Interventions: Other: fNIRS measurement
- Healthy participants at risk: Healthy participants with increased MDD risk (having a 1st-degree relative with MDD)
  Interventions: Other: fNIRS measurement
- Healthy participants low risk: Healthy participants with low MDD risk (having no 1st-degree relatives with MDD)
  Interventions: Other: fNIRS measurement

INTERVENTIONS:
Other: fNIRS measurement — measurement using functional near-infrared spectroscopy

SUMMARY:
Functional near infrared spectroscopy (fNIRS) offers a cheap and reliable tool to investigate prefrontal brain activation in the healthy and diseased human brain. As such, fNIRS bears great potential as a diagnostic tool for clinical practice. Research indicates that fNIRS, together with a relatively simple task to activate the prefrontal cortex, the so-called verbal fluency task (VFT), elucidates prefrontal dysfunction in major depressive disorder (MDD). This finding can potentially serve as an imaging marker for disease pathology, even when depressive symptoms are absent. Indeed, recent research also suggests prefrontal dysfunction in fully remitted MDD (rMDD). Prefrontal haemodynamic responses may therefore serve as a trait marker for MDD vulnerability.

This study aims to investigate the haemodynamic response in rMDD, healthy participants with increased MDD risk (HCr; having a 1st-degree relative with MDD), and low-risk healthy participants (HCnr; having no 1st-degree relatives with MDD) using fNIRS. The investigators hypothesize lower prefrontal reactivity in HCr compared to HCnr, and lowest prefrontal reactivity in rMDD compared to HCnr.

This study has the potential to elucidate the neuronal underpinnings of depression vulnerability in the absence of symptoms that are sometimes considered a confounding factor when it comes to studying the biological encoding of depression.

DETAILED DESCRIPTION:
Healthy participants with a high risk of MDD (HCr), healthy participants with a low risk of MDD (HCnr) and rMDD participants will be included in this study.

Prefrontal haemodynamic response will be measured in all participants during the verbal fluency test (VFT) using 52 channels fNIRS. The VFT involves two neural conditions, one positive condition, and one negative condition.

Both the neuroimage change and the behavioral outcomes of VFT will be compared within-group and among groups. The correlation between the neuroimage change and the behavioral outcomes will be analyzed as well.

ELIGIBILITY:
Inclusion Criteria:

* Mini-mental state examination (MMSE) > 24

Exclusion Criteria:

* Current diagnosis of psychiatric disorders, such as depression, anxiety, schizophrenia, or autism
* current or past diagnosis of neurological disorders, such as head injuries, strokes, encephalitis, epilepsy, Parkinson's, or Alzheimer's

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: rMDD group: People who had major depressive disorders now fully remitted HCr group: Healthy control group with a high risk of depression, refer to as healthy volunteers who have a 1st-degree relative with MDD in this study.
  HCnr group: Healthy control group with a low risk of depression, refer to as healthy volunteers who have no a 1st-degree relative with MDD in this study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Oxygenated hemoglobin (HbO) change during VFT | Up to 6 months
  The HbO change during VFT measuring by fNIRS

SECONDARY OUTCOMES:
Deoxygenated hemoglobin (HbR) change during VFT | Up to 6 months
  The HbR change during VFT measuring by fNIRS
The VFT outcome | Up to 6 months
  The number of correct words during VFT

CONTACTS AND LOCATIONS:
Overall Officials: Georg S Kranz, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong